CLINICAL TRIAL: NCT03890861
Title: Reducing African Americans' Alzheimer's Disease Risk Through Exercise (RAATE)"
Acronym: RAATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Robert L. Newton, Jr., Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2019-002; R01AG062200-01 (NIH)
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Dementia, Alzheimer Type
Keywords: African American; Aging; Physical activity; Cognition; Prevention
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity intervention (Experimental): The intervention group will target 150 minutes of moderate to vigorous aerobic physical activity and two days of strength training, consistent with the current physical activity recommendations. Participants will engage in 2 days per week of supervised activity at community facilities. These participants will be requested to engage in an additional 30 minutes of moderate to vigorous aerobic physical activity two days per week at home.
  Interventions: Behavioral: Physical activity
- Active control (Active Comparator): The active control group will be based on a low-intensity activity program and a healthy aging educational component. The physical activities will include stretching, balance training, flexibility, relaxation, and practicing activities of daily living. The successful aging education component will cover topics including avoiding scams, fall prevention, living wills, and dementia awareness.
  Interventions: Behavioral: Successful Aging

INTERVENTIONS:
Behavioral: Physical activity — Promotion of physical activity to the current federal physical activity guidelines.
  Arms: Physical activity intervention
Behavioral: Successful Aging — Seminars of health topics related to aging in African Americans with light stretching and low intensity activites
  Arms: Active control

SUMMARY:
The RAATE proposal is designed to determine the effects of physical activity on risk factors for Alzheimer's Disease in older African American adults. The study will compare a physical activity program to an active control group. There are three main objectives of the protocol: 1) to determine if a physical activity intervention tailored to older African American adults is effective in modifying cognitive function associated with Alzheimer's Disease, 2) to determine if a physical activity intervention tailored to older African American adults is effective in modifying brain function and structure associated with Alzheimer's Disease, and 3) to determine if a physical activity promotion intervention tailored to African American adults is effective at enhancing physiological parameters. The primary endpoints for the study are episodic memory and executive functioning. The secondary outcomes include anthropometry, blood pressure, brain activation, cerebral blood flow, volume of whole brain and white matter hyperintensities, cardiorespiratory fitness, objectively measured physical activity, circulating hormones, and telomere length.

DETAILED DESCRIPTION:
Alzheimer's disease is steadily increasing in prevalence, with a devastating public health impact. The prevalence of Alzheimer's Disease is higher in African Americans compared to white Americans, thereby constituting a health disparity. Interventions that prevent Alzheimer's disease or change the course of cognitive decline associated with Alzheimer's disease are needed. Most older adults do not achieve recommended levels of physical activity, and this includes African Americans. Regular physical activity has proven to be a safe and effective means to enhance cognitive function in older adults ranging from cognitively healthy to mildly cognitively impaired. Therefore, our study is focused on physical activity promotion, a potent approach to modifying multiple neurobiological pathways implicated in Alzheimer's Disease. We evaluate exercise benefits among elderly African Americans, who are understudied and in whom the natural course of neurodegeneration, exercise effects on neuroprotection and neurodegeneration, and resulting clinical phenotypes may differ. A large body of existing data suggests that exercise improves cardiovascular and cerebrovascular functioning, and thus has the potential to enhance perivascular clearance of amyloid and reduce chronic brain tissue ischemia, among other beneficial effects. At the same time, chronic exercise has been shown to decrease central levels of inflammatory markers and increase central levels of neurotrophic factors, which in turn promote protection against Alzheimer's Disease neurodegeneration pathways via a variety of mechanisms. While physical activity interventions have been shown to have positive effects on these factors and on resultant cognitive functioning in older adults, nearly all interventions have had a negligible representation of African Americans. Prior data suggests that African Americans enter their elderly years against a backdrop of different lifespan exposures to a variety of factors relevant to neuroprotection and neurodegeneration, including cardiovascular risk, exercise, diet, and education. In addition, prior data suggests that the key genetic risk factor for Alzheimer's Disease (APOE) may have differing consequences for Alzheimer's Disease risk among African Americans, and other genetic differences have the potential to influence the brain benefits of physical activity in this community. We will utilize a randomized clinical trial to addresses these questions. Participants will be randomized into a physical activity promotion intervention or a healthy aging information group for 52 weeks. All participants will be of normal cognitive function. We will assess cognitive function, brain structure and function, circulating hormones, objectively measured physical activity, cardiorespiratory fitness, and telomere length. Our study will take the first step toward understanding whether the hypothesized benefits of exercise for the brain carry over to elderly African Americans.

ELIGIBILITY:
Inclusion Criteria:

1. self- identify as African American
2. 60 years and older
3. willing to accept randomization
4. willing to attend group sessions
5. lacking plans to move during the study period
6. free of conditions that would make regular exercise unsafe (e.g. uncontrolled asthma, severe sickle cell disease, etc.)
7. not engaged in regular physical activity
8. Short Physical Performance Battery score >/= 4
9. physically capable of exercise,

Exclusion Criteria:

1. cognitive impairment that would interfere with participating in group interactions
2. unwilling to give written informed consent
3. inability to attend group sessions
4. conditions that prevent regular exercise
5. conditions that the medical or principal investigator determine to warrant exclusion

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2019-08-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in episodic memory | Baseline, 24 weeks, 52 weeks
  The Rey Auditory Verbal Learning Test (RAVLT) is a common neuropsychological tool used to evaluate episodic memory. The RAVLT involves providing participants with 15 unrelated words and asking them to recall the word list. There are 5 trials designed to determine short-term memory and then a 30 minute delay to assess long-term memory. The total words correct in both the short- and long-term trials are used as outcome measures.
Change in executive function | Baseline, 24 weeks, 52 weeks
  The NIH Toolbox Executive Function subdomain consists of the Flanker Inhibitory Control and Attention Test and the Dimensional Change Card Sort Test. The Flanker test is a measure of one's ability to inhibit attention to irrelevant conditions. Participants must identify the direction of a central visual stimuli amongst flanking stimuli either congruent or incongruent with the central stimuli. There are 40 trials and scores range from 0 - 10. The Card Sort is a measure of the ability to shift attention based on rules. Participants must match a target visual stimuli to either a color or word stimuli and this matching shifts during the assessment.

SECONDARY OUTCOMES:
Change in cognitive status | Baseline, 24 weeks, 52 weeks
  The Mini-Mental Status Examination is 30-point questionnaire to assess cognitive impairment.
Change in glucose | Baseline, 24 weeks, 52 weeks
  Fasting levels of glucose will be assessed using standard assays.
Change in time spent in physical activity | Baseline, 24 weeks, 52 weeks
  The Actigraph WGT3X+ accelerometer (ActiGraph LLC, Pensacola, FL) will be worn by the participant for a 7-day period. The device provides both the number of steps per day as well as time in sedentary, light, moderate, and vigorous activity in 1-minute epochs (for adults) using the default filter.
Change in cardiorespiratory fitness | Baseline, 24 weeks, 52 weeks
  All participants will perform a standardized graded exercise testing protocol administered on a treadmill. Fitness will be measured in terms of mL oxygen/kg/min.
Change in physical function-NIH Toolbox | Baseline, 24 weeks, 52 weeks
  Physical function will be assessed using the NIH-TB Motor assessment, which assesses dexterity, balance, locomotion, grip strength, and strength.
Change in telomere length | Baseline, 24 weeks, 52 weeks
  DNA will be extracted from the blood draw and amplified using real-time quantitative polymerase chain reaction (qPCR) to determine average relative telomere length represented by the telomere repeat copy number to single gene copy number (T/S) ratio in triplicate as previously described
Change in weight | Baseline, 24 weeks, 52 weeks
  Weight will be measured using a standard stadiometer. Measurements will be taken to the nearest cm.
Change in brain structure | Baseline, 24 weeks, 52 weeks
  Volumes of the cranial vault, brain tissue, gray matter, white matter, and cerebrospinal fluid, which will be provided as the primary brain structural outcome measures of interest from MRI.
Changes in brain function | Baseline, 24 weeks, 52 weeks
  Pre-selected inhibitory control ROIs (ACC for the Stroop; DLPFC, thalamus, superior frontal, inferior frontal, fusiform, and middle frontal gyri; and ACC and middle frontal gyri for the ANT) are of primary interest.
Change in lipoproteins | Baseline, 24 weeks, 52 weeks
  Fasting levels of lipids will be assessed using standard assays.
APOE genotype | Baseline
  APOE genotype will be assessed using standard assays.
Change in physical activity | Continuously for 52 weeks
  The Fitbit Charge 2 will be worn by participants in both groups.
Change in blood pressure | Blood pressure will be measured using the Omron, Model BP710 automatic blood pressure cuff.
  Blood pressure will be measured using the Omron, Model BP710 automatic blood pressure cuff.
Change in mood | Baseline, 24 weeks, 52 weeks
  The Geriatric Depression Scale will be used to measure depressive symptoms.
Change in height | Baseline, 24 weeks, 52 weeks
  Height will be assessed using a standard stadiometer.
Change in physical function-SPPB | Baseline, 24 weeks, 52 weeks
  Physical function will be assessed using the the Short Physical Performance Battery (SPPB), which is a brief performance battery based on timed short distance walk, repeated chair stands and balance test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Newton, Jr., PhD, Principal Investigator — Pennington Biomedical Research Center; Owen L Carmichael, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
For all study data, Pennington Biomedical has a well-structured internal process for data sharing and transfer. The Office of Legal and Regulatory Compliance is responsible for all data agreements which includes data subject to the protection under HIPAA. As part of the Louisiana State University System, Pennington Biomedical ensures that data agreements are in place in the following circumstances: business associate agreements when the transfer of data contains all identifiers, data use agreements when the transfer of data contains those identifiers that constitute a limited data set and a data transfer agreement in instances where data is de-identified, but still may be subject of protection in order to protect intellectual property rights. Transmission of data to ensure proper safeguards are in place on the data in motion and data at reset are carried out with assistance of the Research Computing Group or the Office of Computing Services.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after data analysis has occurred.